CLINICAL TRIAL: NCT02660788
Title: A Randomised Study of Screening Mammography Return Rates in Overdue Women Due to Standard Screening Mammography Program of British Columbia (Smpbc) Reminders Versus Reminder Letters Signed by Women's Family Physicians
Brief Title: A Randomized Trial of Letters From Family Physicians to Encourage Screening Mammography in Overdue Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: Canadian Breast Cancer Foundation (Other)
Responsible Party: Principal Investigator, Alan Nichol, Radiation Oncologist, British Columbia Cancer Agency
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H12-02832
Record Dates: First submitted 2016-01-18; First posted 2016-01-21 (Estimated); Results first posted 2021-09-02 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Breast Cancer
Keywords: 6-24 months overdue; screening mammography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Arm (Active Comparator): Mail
  Interventions: Other: Standard Reminder Postcard
- Family Physician Reminder Letter Arm (Experimental): Mail
  Interventions: Other: Standard Reminder Postcard; Other: Family Physician Reminder Letter

INTERVENTIONS:
Other: Standard Reminder Postcard
Other: Family Physician Reminder Letter
  Arms: Family Physician Reminder Letter Arm

SUMMARY:
A randomized, double-blinded study conducted in British Columbia, Canada, where there is a publicly funded, organized screening program and screening mammography is recommended at 24-month intervals. Eligible women aged 51-73 years old and overdue for their screening mammogram by 6-24 months are identified in the database of the Screening Mammography Program of BC (SMPBC). Family physicians are recruited by mail and asked to sign letters to the overdue women in their practices. The overdue women are randomized and mailed either the signed reminder letter and the standard reminder postcard, or the standard reminder postcard alone. The primary endpoint is the proportion of overdue women attending a screening mammogram appointment 6 months after the mailing.

ELIGIBILITY:
Inclusion Criteria:

Active family physicians (family physicians, general practitioners or primary care physicians) who have overdue women in their practice that meet the following criteria:

* Previously been enrolled in the SMPBC and had a previous normal screening mammogram.
* Have agreed to being contacted for research on the SMPBC questionnaire
* Are 6-24 months overdue from their last screening mammogram
* Live in BC
* Have listed an active family physician as the contact to receive their mammography results

Exclusion Criteria:

* Family physicians who do not work in primary care
* Family physicians who do not have overdue women in their practice

Ages: 51 Years to 73 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5498 (Actual)
Dates: Start 2013-02; Primary Completion 2013-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Nichol, MD, Principal Investigator — British Columbia Cancer Agency
Locations (1):
- BC Cancer Agency, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chan EK, Wilson C, Tyldesley S, Olivotto IA, Lai A, Sam J, Harry R, Nichol A. Signed family physician reminder letters to women overdue for screening mammography: A randomized clinical trial. J Med Screen. 2018 Sep;25(3):149-154. doi: 10.1177/0969141317719921. Epub 2017 Nov 20. PMID 29157121

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The breast cancer screening program participants were identified by their family physicians
Pre-assignment Details: Only screenees who had not had a mammogram between identification of potential participants and randomization were randomized.
Groups:
- Control Arm: Mail
  Standard Reminder Postcard
- Family Physician Reminder Letter Arm: Mail
  Standard Reminder Postcard
  Family Physician Reminder Letter
Period: Overall Study
Arm/Group | Control Arm | Family Physician Reminder Letter Arm
Started | 2749 | 2749
Completed | 2749 | 2749
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Total includes patients who were screened before randomization
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm | Family Physician Reminder Letter Arm | Total
Number analyzed (Participants) | 2749 | 2749 | 5498
Age, Customized [Number; unit: participants] | 2749 | 2749 | 5498
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2749 | 2749 | 5498
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 2749 | 2749 | 5498

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Overdue Women Returning for Screening Mammography
Description: Percentage of overdue women returning for screening mammography, measured from the date of randomization
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Control Arm | Family Physician Reminder Letter Arm
Number analyzed (Participants) | 2749 | 2749
percentage of participants | 24.0 | 34.4

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Control Arm | Family Physician Reminder Letter Arm
Serious Adverse Events (participants affected / at risk) | 0/2749 | 0/2749
Other Adverse Events (participants affected / at risk) | 0/2749 | 0/2749

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes